CLINICAL TRIAL: NCT04798963
Title: 3D Assessment of Functional Parenchymal Volume and Split Renal Function Before and After Partial Nephrectomy
Brief Title: The Evaluation of Functional Parenchymal Volume and Split Renal Function Before and After Partial Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MACT-PN 2021
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Renal Cell Carcinoma
Keywords: kidney cancer; partial nephrectomy; split renal function
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-clamp partial nephrectomy (Other): Patients who are assigned to on-clamp partial nephrectomy.
  Interventions: Procedure: On-clamp partial nephrectomy
- Off-clamp partial nephrectomy (Other): Patients who are assigned to off-clamp partial nephrectomy.
  Interventions: Procedure: Off-clamp partial nephrectomy

INTERVENTIONS:
Procedure: On-clamp partial nephrectomy — Partial nephrectomy will performed with renal artery clamping (less than or equal to 25 minutes)
  Arms: On-clamp partial nephrectomy
Procedure: Off-clamp partial nephrectomy — Partial nephrectomy will performed without renal artery clamping
  Arms: Off-clamp partial nephrectomy

SUMMARY:
The study aims to compare pre- and postoperative 3D renal function results of patients who underwent on-clamp and off-clamp partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women >18 years; 2. Diagnosis of unilateral renal cell carcinoma (stage T1-T3aN0M0); 3. Planned surgery: retroperitoneoscopic/laparoscopic/robotic partial nephrectomy; 4. Patients with CT of the kidneys with contrast enhancement performed according to the required protocol.

-

Exclusion Criteria:

1. Age < 18 years old or ASA> 3;
2. Solitary kidney;
3. Bilateral kidney
4. The presence of concomitant systemic pathology (DM, AH), as well as kidney disease (glomerulonephritis), which can change the state of the renal parenchyma;
5. Obstructive nephropathy
6. Systemic intake of nephrotoxic drugs;
7. Pregnancy. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-03-02 (Estimated); Study Completion 2022-03-02 (Estimated)

PRIMARY OUTCOMES:
GFR after the surgery | 6 months

SECONDARY OUTCOMES:
Complication rate (Clavien-Dindo) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sechenov University., Moscow, Russia